CLINICAL TRIAL: NCT04131881
Title: The Consistency of Drug Sensitivity in Vitro and Neoadjuvant Chemotherapy Results in Vivo for Early Breast Cancer Patients
Brief Title: The Consistency of Drug Screening in Vitro and Neoadjuvant Chemotherapy Results in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Sponsor
Other Study IDs: PKUPH10B002
Record Dates: First submitted 2019-10-13; First posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer; Drug Effect
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample were retention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neoadjuvant chemotherapy for breast cancer could make unresectable breast cancer be resectable and improve breast conservation rate. Patients with triple negative or Her2 enriched subtype who achieved pCR after neoadjuvant chemotherapy would have better survival. But the overall pCR rate of breast cancer was about 20%. And patients with luminal like subtype were less reactive for neoadjuvant chemotherapy. Improving pCR rate maybe could achieve better survival. So, different methods have tried to select effective drug before chemotherapy.Drug sensitivity screening in vitro for different chemotherapy drugs was a promising method. This study will explore whether drug screening by culturing breast cancer cells in vitro from breast cancer tissue could consistent with neoadjuvant chemotherapy in patients.40 breast cancer patients were recruited.The results of drug sensitivity in vitro and pathological evaluation after neoadjuvant chemotherapy were compared whether they were consistent.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy for breast cancer could make unresectable breast cancer be resectable and improve breast conservation rate. Patients with triple negative or Her2 enriched subtype who achieved pCR after neoadjuvant chemotherapy would have better survival. But the overall pCR rate of breast cancer was about 20%. And patients with luminal like subtype were less reactive for neoadjuvant chemotherapy. Improving pCR rate maybe could achieve better survival. So, different methods have tried to select effective drug before chemotherapy.Drug sensitivity screening in vitro for different chemotherapy drugs was a promising method. This study will explore whether drug screening by culturing breast cancer cells in vitro from breast cancer tissue could consistent with neoadjuvant chemotherapy in patients.40 breast cancer patients who would receive neoadjuvant chemotherapy were recruited.Breast cancer tissues were obtained before chemotherapy. The breast cancer cells were cultured in unadhesive dishes. Chemotherapy drugs were put in dishes and drug sensitivity were evaluated. Patients received operation and pathological evaluationc after neoadjuvant chemotherapy. The results of drug sensitivity in vitro and pathological evaluation after neoadjuvant chemotherapy were compared whether they were consistent.

ELIGIBILITY:
Inclusion Criteria:

* invasive breast cancer candidates for neoadjuvant chemotherapy agreed to participate in this observative experiments could receive operation normal liver and renal function

Exclusion Criteria:

* inflammatory breast cancer recurrent breast cancer

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in this study were invasive early breast cancer patients who were candidate for neoadjuvant chemotherapy.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Consistency rate of drug sensitivity in vitro and in vivo | through study completion, an average of 2 years
  Compute the percentage of patients whose drug sensitivity were consistent between in vitro and in vivo, as both were sensitive or insensitive.

CONTACTS AND LOCATIONS:
Overall Officials: Shu Wang, doctor, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People'S Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No